CLINICAL TRIAL: NCT06488313
Title: A Phase 2a, Open-label, Multiple Ascending Dose Study to Evaluate the Pharmacodynamics and Safety of ARCT-810 in Adolescent and Adult Participants With Ornithine Transcarbamylase Deficiency
Brief Title: A Study to Evaluate the Pharmacodynamics and Safety of ARCT-810 in Participants With OTCD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arcturus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARCT-810-04
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: OTC Deficiency; Ornithine Transcarbamylase Deficiency; OTCD
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Intervention Model Description: All participants will receive 5 doses of Study Drug via intravenous infusion at one of the three dose levels. Dose levels will be enrolled sequentially.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARCT-810 (Experimental): Participants will receive up to 5 IV infusions of ARCT-810 administered at 14-day intervals.
  Interventions: Biological: ARCT-810

INTERVENTIONS:
Biological: ARCT-810 — ARCT-810 is an investigational medicinal product comprising Ornithine Transcarbamylase (OTC) messenger RNA (mRNA) formulated in a lipid nanoparticle (LNP).

SUMMARY:
Evaluate the safety and pharmacodynamics of multiple doses of ARCT-810 in adolescent and adult participants with OTC deficiency.

DETAILED DESCRIPTION:
This a Phase 2a, open-label study of ARCT-810 in participants 12 years of age and older living with OTC deficiency. After a diet stabilization period of at least 4 weeks, all participants will be enrolled to receive ARCT-810 every two weeks, for up to five doses, at one of three dose levels. Clinic visits will occur during screening and at Days 1, 15, 29, 36, 43, 57, 60, 71, and 85. During the study, participants will remain on their current clinical management for OTC deficiency. Dose escalation or cohort expansion may occur following completion of three participants at each dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to comply with all the protocol requirements, complete all study visits and sign informed consent.
2. Males and Females aged ≥12 years, at Screening.
3. Documented clinical diagnosis of OTC deficiency.
4. History of symptomatic hyperammonemia or elevated plasma ammonia or glutamine with clinical stability for at least 1 month prior to Screening.
5. Medically managed for OTC deficiency and receiving a stable protein-restricted diet, dietary supplements, and/or ammonia scavenger regimen (if applicable) for at least 28 days.
6. Good general health with no clinically significant abnormal findings that would interfere with study procedures (including plasma ammonia within participant's historical range).
7. Must be willing to adhere to contraception guidelines.

Exclusion Criteria:

1. Uncontrolled hypertension.
2. Symptoms of infection for at least 7 days prior to dosing.
3. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
4. History of any OTC gene therapy, or history of liver-derived stem cell therapy in the past 2 years.
5. History of any organ transplant.
6. History of severe allergic reaction to a liposomal or PEG-containing product.
7. History of congenital or acquired cardiac disorders.
8. Abuse of medications, illicit drugs or alcohol.
9. Blood donation of 50 to 499 mL within 30 days of screening or of >499 mL within 60 days of screening.
10. Clinically significant laboratory abnormalities on screening labs including INR >1.5, eGFR< 60 mL/min/1.73m2 or positive test results for HIV, HBV, or HCV.
11. Inadequately controlled diabetes.
12. Clinically significant anemia.
13. Changes in maintenance therapies for OTC deficiency with 28 days prior to dosing.
14. Medical history requiring continuous or intermittent systemic corticosteroid administration.
15. Receipt of inhibitors of urea synthesis or drugs that significantly affect renal clearance.
16. Recent treatment with another investigational drug, biological agent, or device.
17. Treatment with any oligonucleotide (siRNA or mRNA) within 6 months prior to screening. COVID-19 vaccines are not exclusionary.
18. Involved in study conduct or an immediate family member of an individual involved in the study.
19. Participated in another dosing cohort of the study.
20. Any other conditions, in the opinion of the investigator, that would interfere with participation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and dose-relationship of adverse events (AEs) | Day 85
  Safety and tolerability of ARCT-810 assessed by incidence, severity, and dose-relationship of AEs

SECONDARY OUTCOMES:
Stable isotope ureagenesis assay values (AUC of first isotope) | Up to Day 85
  Change from Baseline in stable isotope ureagenesis assay values (AUC of first isotope) following multiple doses of ARCT-810
Stable isotope ureagenesis assay values (AUC of second isotope) | Up to Day 85
  Change from Baseline in stable isotope ureagenesis assay values (AUC of second isotope) following mulitple doses of ARCT-810
Fasting plasma ammonia | Up to Day 85
  Proportion of participants maintaining normal morning fasting plasma ammonia
Plasma Glutamine | Up to Day 85
  Change from Baseline in plasma glutamine and labeled glutamine as available
Plasma pharmacokinetics | Up to Day 57
  The noncompartmental plasma pharmacokinetics of ARCT-810 will be assessed based on the observed plasma concentration of ARCT-810 mRNA and lipid

CONTACTS AND LOCATIONS:
Locations (1):
- Uncommon Cures, Chevy Chase, Maryland, United States

IPD SHARING:
Plan to Share IPD: No